CLINICAL TRIAL: NCT00144703
Title: Open Label Phase II Trial of Sirolimus in Combination With Tacrolimus for Graft-vs-Host Disease Prophylaxis After Matched, Related Allogeneic Hematopoietic Stem Cell Transplantation
Brief Title: Sirolimus With Tacrolimus for Graft-vs-Host Disease Prophylaxis After Related Stem Cell Transplantation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Corey S. Cutler, MD, MPH, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 02-090
Record Dates: First submitted 2005-09-01; First posted 2005-09-05 (Estimated); Last update posted 2012-01-26 (Estimated); Status verified 2009-01

CONDITIONS: Hematologic Malignancies; Myelogenous Leukemia; Acute Lymphoblastic Leukemia; Myelodysplastic Syndrome; Non-Hodgkin's Lymphoma; Hodgkin's Disease
Keywords: Graft versus host disease; GVHD; Stem cell transplantation; sirolimus; tacrolimus
MeSH Terms: conditions — Hematologic Neoplasms; Leukemia, Myeloid; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Myelodysplastic Syndromes; Lymphoma, Non-Hodgkin; Hodgkin Disease; Graft vs Host Disease | interventions — Sirolimus; Tacrolimus

INTERVENTIONS:
Drug: Sirolimus
Drug: Tacrolimus

SUMMARY:
The purpose of this study is to evaluate the ability of sirolimus to prevent graft versus host disease (GVHD) in patients following stem cell transplant from a related donor.

DETAILED DESCRIPTION:
* Therapy to prevent GVHD will consist of an infusion of tacrolimus intravenously and sirolimus orally once per day starting 3 days before stem cell infusion. This will take place in the hospital where the patient will remain for the duration of the transplant.
* Sirolimus will continue for 9 weeks at at stable dose, then will be tapered by 1/3 on week 9 and 1/3 on week 17. It will be stopped on week 26 if there is no significant evidence of GVHD. These dose modifications will occur at home and patients will be seen weekly for the first 2 months after discharge.
* If GVHD is present, the tapering schedule wil be slower and based upon the patient's clinical condition.
* Tacrolimus will be given orally once the patient is discharged from the hospital and will be tapered at the same schedule as sirolimus. Blood levels of both tacrolimus and sirolimus will be monitored and the dose adjusted accordingly.
* During the year following stem cell transplant, blood work will be performed to evaluate the immune system and GVHD.

ELIGIBILITY:
Inclusion Criteria:

* Patients with hematologic malignancies who will undergo allogeneic HSCT from matched family-members.
* Age greater than 18
* ECOG performance status 0-2
* Total bilirubin < 2.0 mg/dl
* AST < 90 IU
* Serum creatinine < 2.0 mg/dl

Exclusion Criteria:

* Active, uncontrolled infection
* Ejection fraction < 45% by echocardiogram or MUGA scan
* Forced vital capacity < 60%
* Uncontrolled hypertension
* Second transplantation
* Evidence of HIV infection
* Cholesterol > 300 mg/dl
* Relapsed aggressive Burkitt's or Burkitt's-like lymphoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55
Dates: Start 2002-07; Primary Completion 2006-11 (Actual); Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
To determine the feasibility of using sirolimus and tacrolimus without methotrexate for GVHD prophylaxis after stem cell transplantation.

SECONDARY OUTCOMES:
To compare the rates of grade II-IV and III-IV acute GVHD with historical controls
to determine the incidence of 100 day mortality after stem cell transplant using this regimen
to determine the overall survival at 1 year after transplantation in this patient population.

CONTACTS AND LOCATIONS:
Overall Officials: Corey Cutler, MD, MPH, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana-Farber Cancer Institute, Boston, Massachusetts, United States